## Adjuvant Radiotherapy for Resected Hepatocellular Carcinoma With MVI

NCT 04891874 2015-8-1

## Statistical analysis

The comparison of clinical parameters between the two groups were conducted by the Student's t test, the Mann Whitney U-test, the Chi-square test or Fisher's exact test, relying on the variables as appropriate. The DFS and OS were determined by the Kaplan-Meier method which was generated by the log-rank test. The univariate and multivariate analyses were conducted to identify the independent risk factors of DFS and OS in the entire group of BCLC 0/A patients receiving operation in the recruitment period. Variables with P < 0.1 on univariable analysis were subjected to the multivariable Cox regression model using a forward stepwise variable selection. The statistical significance level was set at P < 0.05 in all the analyses.